CLINICAL TRIAL: NCT04530500
Title: In-vitro Diagnostic Test to Predict COVID-19 Mortality and Disease Severity
Brief Title: COVID-19 In-vitro Diagnostic Test and Androgen Receptor Gene Expression
Status: Withdrawn | Type: Observational
Why Stopped: Covid pandemic prohibited us from completing study-related activities.
Sponsor: University of California, Irvine (Other)
Collaborators: Applied Biology, Inc. (Industry)
Responsible Party: Principal Investigator, Natasha Mesinkovska, Director of Clinical Research, University of California, Irvine
Other Study IDs: 20205907
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Covid19; Androgen Receptor Gene Overexpression
Keywords: androgen receptor; severity; mortality
MeSH Terms: conditions — COVID-19; Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Arm 1: Males first tested positive for SARS-CoV-2 at the site (medical center) with CAG length <24 (based on the CoVAST Test)
  Interventions: Genetic: COVID-19 Androgen Sensitivity Test (CoVAST)
- Arm 2: Males first tested for SARS-CoV-2 at the site (medical center) with CAG length >=24 (based on the CoVAST Test)
  Interventions: Genetic: COVID-19 Androgen Sensitivity Test (CoVAST)

INTERVENTIONS:
Genetic: COVID-19 Androgen Sensitivity Test (CoVAST) — The CoVAST Test is an in-vitro non diagnostic test. The test reports the genetic health risk of male patients in developing severe symptoms following COVID 19 infection. The genetic information provided by this test will help physicians evaluate the association of AR gene polymorphism with disease severity and mortality following COVID-19 infection. The CoVAST Test is indicated for reporting of the following variant associated with the following gene.

SUMMARY:
This research study will evaluate the association of Androgen Receptor (AR) gene expression and COVID-19 disease severity and mortality. The research procedure involves collection of a single saliva sample which will be mailed to the participants by the study team. This saliva will be used in a COVID-19 Androgen Sensitivity Test (CoVAST) which will detect AR gene expression. Eligible participants are males, at least 18 years or older, and have tested positive for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Male over the age of 18
* Laboratory confirmed SARS-CoV-2 infection
* Able to give verbal informed consent

Exclusion Criteria:

* Unable to give informed consent
* Diagnosed with an additional respiratory co-infection
* XXY males

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males over age 18 who have tested positive for SARS-CoV-2 infection within the University of California, Irvine Health System.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients deceased | 28 days
  Number of subjects deceased at or before 28 days

SECONDARY OUTCOMES:
Number of patients discharged | 14 days
  Number of patients discharged at or before 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Mesinkovska, MD, PhD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Applied Biology, Inc, Irvine, California
  - University of California, Irvine - Dermatology Clinical Research, Irvine, California

IPD SHARING:
Plan to Share IPD: No